CLINICAL TRIAL: NCT03661086
Title: Oxygen Control and Weaning by O2matic to Patients Admitted With an Exacerbation of COPD
Acronym: O2MATIC-WEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Ejvind Frausing Hansen, Senior Consultant, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O2MATIC-O2WEAN
Record Dates: First submitted 2018-09-01; First posted 2018-09-07 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: COPD Exacerbation; Hypoxia; Hypoxemia; Hyperoxia; Respiratory Failure; Respiratory Insufficiency; Copd Exacerbation Acute
Keywords: closed-loop; oxygen treatment
MeSH Terms: conditions — Hypoxia; Hyperoxia; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled parallel study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- O2matic (Active Comparator): Usual care plus O2matic controlled oxygen therapy for a maximum of 3 days or until weaning from oxygen supplementation
  Interventions: Device: O2matic
- Manual (No Intervention): Usual care plus manual controlled oxygen therapy by nursing staff. O2matic used in monitoring mode to measure SpO2 continuously.

INTERVENTIONS:
Device: O2matic — O2matic controls oxygen with the aim of maintaining SpO2 within a predefined target interval, e.g. 88-92 % with the lowest possible supplementation of oxygen by nasal cannula
  Arms: O2matic

SUMMARY:
The aim of the study is to examine if automated oxygen delivery with O2matic allows for faster weaning from oxygen and better oxygen control than manually controlled oxygen therapy for patients admitted with an exacerbation of chronic obstructive pulmonary disease (COPD). Furthermore it will be tested if O2matic compared to manual control allows for faster discharge from hospital. Patients sense of security, anxiety and dyspnea will be evaluated by questionnaires.

DETAILED DESCRIPTION:
Closed-loop control of oxygen therapy is described in the literature used for preterm infants, trauma patients, medical emergency use and patients with COPD. For the latter, closed-loop therapy has been used for patients admitted to hospital with an exacerbation, for domiciliary oxygen use and during exercise. O2matic is a closed-loop system that is based on continuous and non-invasive measurement of pulse and oxygen-saturation (SpO2). The algorithm in O2matic controls oxygen delivery with the aim of keeping the SpO2 within the desired interval, which could be 88-92 % for COPD-patients in accordance with international guidelines on this topic. SpO2-interval can be set for the individual patients, as can the range of acceptable oxygen-flow. If SpO2 or oxygen-flow cannot be maintained within the desired intervals an alarm will sound.

All studies on closed-loop systems have shown that this method is better than manually control by nurse to maintain saturation within the desired interval. Furthermore, some studies have indicated that closed-loop has the possibility to reduce admission time and to reduce time spent with oxygen therapy, due to more efficient and fast withdrawal from oxygen supplementation.

In the present study O2matic will be tested versus manual control, for patients admitted with an exacerbation in COPD, and in need of supplemental oxygen. During the study the patients will either have oxygen controlled with O2matic or manually by nursing staff for 3 consecutive days. All patients will have continuous logging of pulse, oxygen-saturation and oxygen-flow with O2matic, but only in the O2matic active group, the algorithm will control oxygen-delivery.

The primary hypothesis is that O2matic compared to manual control allows for faster weaning from oxygen supplementation, and that more patients will be weaned from oxygen supplementation within a time frame of 3 days. Furthermore it will be tested if O2matic compared to manual control leads to faster achieved respiratory stability, allowing for hospital discharge. It will be tested if O2matic is better than manual control in maintaining oxygen-saturation within the desired interval and reducing time with unintended hypoxia and hyperoxia. Patients sense of security and feeling of anxiety and dyspnea will be evaluated by questionnaires.

No safety issues has been reported in the literature. O2matic is approved for clinical testing by The Danish Medicines Agency, The Ethics Committee in the Capital Region of Denmark and by the regional Data Protection Board. The study will be conducted according to Good Clinical Practice (GCP) standards with independent monitoring. All adverse events and serious adverse events will be monitored and serious adverse events will be reported to Danish Medicines Agency.

ELIGIBILITY:
Inclusion Criteria:

* COPD verified by Forced Expiratory Volume in 1. second (FEV1) divided by Forced Vital Capacity (FVC) < 0,70
* Admission due to exacerbation in COPD
* COPD exacerbation and pneumonia can be included
* Expected duration of admission > 48 hours
* Need for oxygen supplementation (SpO2 <= 88 % on room air)
* Cognitively able to participate in the study
* Willing to participate and give informed consent

Exclusion Criteria:

* Need or anticipated need for mechanical ventilation (intermittent Continuous Positive Airway Pressure (CPAP) is allowed)
* Major comorbidities causing hypoxemia (Cancer, heart disease, pulmonary emboli)
* Asthma or other respiratory condition requiring higher SpO2 than normal for COPD
* Pregnancy
* Cognitive barriers for participation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Time to weaning from oxygen supplementation | 30 days
  Time to weaning from oxygen supplementation in O2matic and manual arm (Patients will be followed for this outcome during the admission, up to 30 days)

SECONDARY OUTCOMES:
Number of patients weaned from oxygen supplementation after day 1 | 1 day
  Fraction of patients weaned from oxygen supplementation after 1 day in O2matic and manual arm
Number of patients weaned from oxygen supplementation after day 3 | 3 days
  Fraction of patients weaned from oxygen supplementation after 3 days in O2matic and manual arm
Time within SpO2 interval | 3 days
  Fraction of time within prescribed SpO2 interval in O2matic and manual arm
Time with severe hypoxemia | 3 days
  Fraction of time with SpO2 < 85 % in O2matic and manual arm
Time with minor hypoxemia | 3 days
  Fraction of time with SpO2 below target but not below 85 % in O2matic and manual arm
Time with hyperoxia | 3 days
  Fraction of time with SpO2 above target in O2matic and manual arm
Sensation of safety | 3 days
  Patients sensation of safety measured by Visual Analog Scale (VAS) score in O2matic and manual arm
Sensation of anxiety | 3 days
  Patients sensation of anxiety measured by Hospital Anxiety and Depression (HADS-A ) subscale in O2matic and manual arm
Sensation of dyspnea | 3 days
  Patients sensation of dyspnea measured by Multidimensional Dyspnea Profile (MDP) in O2matic and manual arm
Time to discharge | 30 days
  Time from admission to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Vestbo, DMSc, Study Chair — Manchester University Hospital
Locations (5):
- Denmark (5):
  - Bispebjerg University Hospital, Copenhagen
  - Nordsjællands Hospital, Frederikssund
  - Gentofte University Hospital, Hellerup
  - Herlev University Hospital, Herlev
  - Hvidovre University Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rice KL, Schmidt MF, Buan JS, Lebahn F, Schwarzock TK. AccuO2 oximetry-driven oxygen-conserving device versus fixed-dose oxygen devices in stable COPD patients. Respir Care. 2011 Dec;56(12):1901-5. PMID 22288082
- [Background] Cirio S, Nava S. Pilot study of a new device to titrate oxygen flow in hypoxic patients on long-term oxygen therapy. Respir Care. 2011 Apr;56(4):429-34. doi: 10.4187/respcare.00983. Epub 2011 Jan 21. PMID 21255511
- [Background] Lellouche F, L'her E. Automated oxygen flow titration to maintain constant oxygenation. Respir Care. 2012 Aug;57(8):1254-62. doi: 10.4187/respcare.01343. Epub 2012 Feb 17. PMID 22348812
- [Background] Lellouche F, Bouchard PA, Roberge M, Simard S, L'Her E, Maltais F, Lacasse Y. Automated oxygen titration and weaning with FreeO2 in patients with acute exacerbation of COPD: a pilot randomized trial. Int J Chron Obstruct Pulmon Dis. 2016 Aug 24;11:1983-90. doi: 10.2147/COPD.S112820. eCollection 2016. PMID 27601891
- [Background] Lellouche F, L'Her E, Bouchard PA, Brouillard C, Maltais F. Automatic Oxygen Titration During Walking in Subjects With COPD: A Randomized Crossover Controlled Study. Respir Care. 2016 Nov;61(11):1456-1464. doi: 10.4187/respcare.04406. Epub 2016 Oct 18. PMID 27794080
- [Background] L'Her E, Dias P, Gouillou M, Riou A, Souquiere L, Paleiron N, Archambault P, Bouchard PA, Lellouche F. Automatic versus manual oxygen administration in the emergency department. Eur Respir J. 2017 Jul 20;50(1):1602552. doi: 10.1183/13993003.02552-2016. Print 2017 Jul. PMID 28729473
- [Background] Hansen EF, Hove JD, Bech CS, Jensen JS, Kallemose T, Vestbo J. Automated oxygen control with O2matic(R) during admission with exacerbation of COPD. Int J Chron Obstruct Pulmon Dis. 2018 Dec 14;13:3997-4003. doi: 10.2147/COPD.S183762. eCollection 2018. PMID 30587955
- See also: Background and description of the O2matic device — http://O2matic.com